CLINICAL TRIAL: NCT00481780
Title: Conventional Balloon Angioplasty vs. Cutting Balloon Angioplasty for Treatment of Femoropopliteal Artery In-Stent Restenosis - A Randomized Controlled Pilot Trial
Brief Title: PTA vs. CB-PTA for Treatment of Femoropopliteal Artery In-Stent Restenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-05

CONDITIONS: Instent Restenosis; Cutting Balloon Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: plain balloon angioplasty
Device: cutting balloon angioplasty

SUMMARY:
Percutaneous transluminal angioplasty (PTA) is a minimally invasive technique for treatment of superficial femoropopliteal artery (SFA) obstructions or occlusions in patients with intermittent claudication as well as critical limb ischemia. Initial technical success rates of above 95% can be achieved and acceptably low rates of complications are consistently reported in the literature. There is a direct relation between treated vessel length and patency rates. One year patency of lesions longer than 10cm has only been 22% at one-year follow up. This major drawback limits a widespread applicability of PTA, and the indication of PTA particularly in patients with intermittent claudication is discussed controversially.With the introduction of endovascular stents, the problems of elastic recoil and residual stenoses due to arterial dissection could be resolved and initial reports of stenting for the treatment of occlusive atherosclerotic disease of the SFA showed promising results with primary and secondary patency rates of 87% to 90% after 18 months. However, subsequent studies demonstrated that exaggerated neo-intimal hyperplasia in the stented segment frequently leads to instent restenosis. This condition will be of greater importance with increasing number of stent implantation procedures during the last years. The concept of cutting balloon seems appealing for this indication, as the balloon-mounted microtomes guarantee smooth lumen gain within the stent, without the risk of vessel wall perforation. Initial reports of the use of the cutting balloon for the treatment of occlusive atherosclerotic disease of the SFA show promising results, indicating that the problems of elastic recoil and residual stenoses due to arterial dissection might be resolved. The cutting balloon has four tiny microtomes (< 0.1mm height) on the outside, which cut the fibrous plaque during expansion of the balloon. Consequently the problem of elastic recoil is ideally addressed, additionally less trauma is exercised on the vessel wall during dilatation of the balloon. This might be achieved by a reduction of vessel wall trauma, vessel wall inflammation and consequently reduced neointimal formation. Although the indications for CB-PTA in the SFA includes significant residual stenosis or in-stent restenosis, there are currently no published randomized controlled trials (RCT) comparing PTA vs. cutting balloon angioplasty (CB-PTA) for any specific condition. This lack of data led us to initiate a RCT comparing primary PTA vs. CB-PTA for treatment of in-stent restenoses in patients with intermittent claudication or critical limb ischemia with TASC category A-B in the femoropopliteal artery .

DETAILED DESCRIPTION:
Percutaneous transluminal angioplasty (PTA) is a minimally invasive technique for treatment of superficial femoropopliteal artery (SFA) obstructions or occlusions in patients with intermittent claudication as well as critical limb ischemia. Initial technical success rates of above 95% can be achieved and acceptably low rates of complications are consistently reported in the literature. There is a direct relation between treated vessel length and patency rates. One year patency of lesions longer than 10cm has only been 22% at one-year follow up. This major drawback limits a widespread applicability of PTA, and the indication of PTA particularly in patients with intermittent claudication is discussed controversially.

With the introduction of endovascular stents, the problems of elastic recoil and residual stenoses due to arterial dissection could be resolved and initial reports of stenting for the treatment of occlusive atherosclerotic disease of the SFA showed promising results with primary and secondary patency rates of 87% to 90% after 18 months. However, subsequent studies demonstrated that exaggerated neo-intimal hyperplasia in the stented segment frequently leads to instent restenosis. This condition will be of greater importance with increasing number of stent implantation procedures during the last years. Repeated PTA of instent restenosis is performed for revascularisation in these patients, but the gold standard for treatment of instent restenosis is unknown and the rate of recurrence after repeat treatment of instent restenosis remains high. The concept of cutting balloon seems appealing for this indication, as the balloon-mounted microtomes guarantee smooth lumen gain within the stent, without the risk of vessel wall perforation (due to the protecting effect of the stent as the outer limit for the microtomes).

Initial reports of the use of the cutting balloon for the treatment of occlusive atherosclerotic disease of the SFA show promising results, indicating that the problems of elastic recoil and residual stenoses due to arterial dissection might be resolved. The cutting balloon has four tiny microtomes (< 0.1mm height) on the outside, which cut the fibrous plaque during expansion of the balloon. Consequently the problem of elastic recoil is ideally addressed, additionally less trauma is exercised on the vessel wall during dilatation of the balloon. This might be achieved by a reduction of vessel wall trauma, vessel wall inflammation and consequently reduced neointimal formation. The cutting balloon can be used for pre-dilatation with diameters slightly less than the target vessel diameter, but still cuts the fibrous plaque, the desired target vessel diameter is then achieved by final touch up dilatation with a standard angioplasty balloon. In the coronary arteries the cutting balloon has been used in randomized studies comparing CB-PTCA to PTCA, as well as in trials for the treatment of in-stent restenosis. All of these trials demonstrated the safety and efficacy of the cutting balloon, only larger randomized trials failed to proof superiority to conventional PTCA. Data in the peripheral arteries are at least scarce. Although the indications for CB-PTA in the SFA includes significant residual stenosis or in-stent restenosis, there are currently no published randomized controlled trials (RCT) comparing PTA vs. cutting balloon angioplasty (CB-PTA) for any specific condition. This lack of data led us to initiate a RCT comparing primary PTA vs. CB-PTA for treatment of in-stent restenoses in patients with intermittent claudication or critical limb ischemia with TASC category A-B in the femoropopliteal artery . The primary endpoint is the occurrence of restenosis as an ultrasonographic reduction of the vessel lumen diameter >50% within 6 months after endovascular treatment. In addition, the course of postintervention inflammation as indicated by serum levels of C-reactive protein (CRP), serum amyloid A (SAA) and fibrinogen will be assessed.

STUDY DESIGN, INCLUSION AND EXCLUSION CRITERIA. Patients with in-stent restenosis (ultrasonographic stenosis > 50% of the vessel lumen diameter) after prior PTA and Stent placement of the SFA will be enrolled to this single-center prospective RCT. The protocol has to be approved by the institutional ethics committee and all patients have to provide written informed consent before enrollment. Entry criteria include symptomatic peripheral artery disease with intermittent claudication (Fontaine stage IIa or b), or critical limb ischemia related to a recurrent stenosis in a previously stented segment of up to 20 cm length. Exclusion criteria history of intolerance of anti-platelet therapy, or adverse reaction to heparin, bleeding diathesis, creatinine >2.5 mg/dL, hemodialysis, active bacterial infection, and allergy to contrast media, pregnancy and disability to give informed consent.

FOLLOW-UP. ABI testing, treadmill exercise, and Duplex-sonography of the treated vessels will be performed in all patients at 1, 3, and 6 months after treatment. A peak systolic velocity of ≥ 2.4 was considered indicative of a >50% narrowing and was defined as indicative of a restenosis10. Reintervention or surgical bypass at the treated segment are also defined as a restenosis and loss of primary patency. An improvement of at least one Fontaine category above baseline is used to define clinical success in association with maintenance of at least a 0.15 increase in exercise ABI from the preprocedure level.

COMPLICATIONS are classified as either major or minor (as described in Appendix A). Major complications are e.g. bleedings at the puncture side with hematoma and a decrease of serum hemoglobin more than 2 g/dl, loss of stent in the artery , vessel rupture, amputation, macroembolisation with need for further revascularisation and life threatening bleeding complications.

STUDY ENDPOINTS. The primary study endpoint is the occurrence of a >50% restenosis at the treated segment at 6 months post-intervention as determined by duplex ultrasound (in-segment restenosis). Secondary objectives are primary technical success rates (residual stenosis <30% without need for secondary stent implantation, primary assisted and secondary patency, clinical patency, target vessel and target lesion revascularization, and cardiovascular adverse events at 1, 3, and 6 months after the procedure. Furthermore, the course of inflammatory parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients with in-stent restenosis (ultrasonographic stenosis > 50% of the vessel lumen diameter) after prior PTA and Stent placement of the SFA
* symptomatic peripheral artery disease with intermittent claudication or critical limb ischemia

Exclusion Criteria:

* history of intolerance of anti-platelet therapy
* adverse reaction to heparin
* bleeding diathesis
* creatinine >2.5 mg/dL
* hemodialysis
* active bacterial infection
* allergy to contrast media
* pregnancy
* disability to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-11; Study Completion 2007-04

PRIMARY OUTCOMES:
The primary study endpoint is the occurrence of a >50% restenosis at the treated segment at 6 months postintervention as determined by duplex ultrasound (in-segment restenosis) | within 6 months follow up

SECONDARY OUTCOMES:
primary technical success rates residual stenosis <30% without need for secondary stent implantation, primary assisted and secondary patency, clinical patency, target vessel and target lesion revascularization, cardiovascular adverse events | within 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Minar Erich, Prof.Dr., Principal Investigator — General Hospital of Vienna
Locations (1):
- General Hospital of Vienna, Vienna, Austria